CLINICAL TRIAL: NCT01397175
Title: A Multicenter, Open-labeled, Randomized Controlled Trial Comparing Three 2nd Generation Drug-Eluting Stents in Real-World Practice
Brief Title: BES, EES, and ZES-R in Real World Practice
Acronym: CHOICE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow enrollment
Sponsor: Yonsei University (Other)
Collaborators: Gangwon Cardiovascular Health Research Institute (Other)
Responsible Party: Principal Investigator, Yoon Junghan, Professor of Cardiology, Department of Internal Medicine, Yonsei University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHOICE
Record Dates: First submitted 2011-07-05; First posted 2011-07-19 (Estimated); Last update posted 2019-07-09 (Actual); Status verified 2019-07

CONDITIONS: Coronary Artery Disease
Keywords: Coronary artery disease; Percutaneous coronary intervention; Drug-eluting stent
MeSH Terms: conditions — Coronary Artery Disease | interventions — Biosensing Techniques

STUDY DESIGN:
Intervention Model Description: BES EES ZES-R
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Biolimus-eluting stent (Active Comparator): Biomatrix stent, Biosensors, USA Biomatrix Flex stent, Biosensors, USA
  Interventions: Device: Biolimus-eluting stent
- Everolimus-eluting stent (Active Comparator): Xience Prime stent, Abbott, USA Xience V stent, Abbott, USA
  Interventions: Device: Everolimus-eluting stent
- Zotarolimus-eluting stent (Active Comparator): Endeavor resolute, Medtronic, USA Endeavor resolute integrity, Medtronic, USA
  Interventions: Device: Zotarolimus-eluting stent

INTERVENTIONS:
Device: Biolimus-eluting stent — Biolimus-eluting stent (BES, BioMatrix or BioMatrix Flex, Biosensors, USA) has bio-degradable polymer which is consisted with poly-lactic acid (PLA) and degraded into H2O and CO2 while releasing the biolimus. BES would be expected to reduce the stent thrombosis comparing with the DES with durable polymer.
  Other Names: Biomatrix, Biosensors, USA; Biomatrix flex, Biosensors, USA
  Arms: Biolimus-eluting stent
Device: Everolimus-eluting stent — Everolimus-eluting stent (EES, Xience V or Xience Prime, Abbott, USA) use the MULTILINK VISION stent platform and durable polymer containing everolimus. It has the thinnest strut thickness among the available DES in Korea.
  Other Names: Xience V, Abbott, USA; Xience Prime, Abbott, USA
  Arms: Everolimus-eluting stent
Device: Zotarolimus-eluting stent — Zotarolimus-eluting stent with biolinx polymer (ZES, Endeavor Resolute or Endeavor Resolute Intergrity, Medtronic, USA) has DRIVER stent platform. The durable polymer in this DES has changed from phosphorylcholine (PC) polymer which was used in Endeavor to Biolinx polymer which has more biocompatible features.
  Other Names: Endeavor Resolute, Medtronic, USA; Endeavor Resolute Integrity, Medtronic, USA
  Arms: Zotarolimus-eluting stent

SUMMARY:
The primary objective of this study is to compare the rate of device-oriented composite consisted of cardiac death, myocardial infarction not clearly attributable to a nontarget vessel, and clinically indicated target lesion revascularization among the patients treated with EES, ZES-R, or BES at 24-month clinical follow-up post-index procedure. Trial end points are summarized in Table I. The hypothesis is that BES is equivalent to EES or BES is equivalent to ZES-R at the primary end point.

DETAILED DESCRIPTION:
Previous randomized trials have shown the superior efficacy of drug-eluting stents (DES), such as sirolimus-eluting stent (SES, CYPHER, Cordis, US), paclitaxel-eluting stent (PES, TAXUS, Boston Scientific, US), and zotarolimus-eluting stent (ZES, Endeavor, Medtronic, US) compared with bare metal stents (BMS) by reducing neointimal hyperplasia, late luminal loss, and angiographic restenosis leading to decreased target lesion revascularization. Unfortunately, restenosis still occurs and late stent thrombosis can develop by delaying endoluminal healing or by chronic inflammation.Accordingly, development of new DES is required to improve efficacy by reducing revascularization and safety by reducing the risk of stent thrombosis. With the improvement of polymer, drug, and the platform, the 2nd generation DES, including everolimus-eluting stent (EES, Xience V or Xience Prime, Abbott, USA), zotarolimus-eluting stent with biolinx polymer (ZES-R, Endeavor Resolute or Endeavor Resolute Integrity, Medtronic, USA), and biolimus-eluting stent (BES, BioMatrix or Biomatrix Flex, Biosensors, USA), have been shown to be superior or non-inferior in safety and efficacy trials compared with 1st generation DES.

However, it is difficult to know if there are any differences in efficacy and safety between the EES, the ZES-R, and the BES, in real world practice due to the lack of data comparing these three 2nd generation DES directly. This study provides the evidence for the CHOICE of stent when physicians are treating patients by percutaneous coronary intervention.

ELIGIBILITY:
Inclusion Criteria

* Age > 19 years
* Subject is able to verbally confirm understanding of risks, benefits and treatment alternatives of receiving the drug-eluting stent(s) and he/she or his/her legally authorized representative provides written informed consent prior to any study related procedure
* Subject must have significant stenosis (>50% by visual estimate) on a native or in-stent coronary artery
* Subject must have evidence of myocardial ischemia (e.g., stable, unstable angina, recent infarction, acute myocardial infarction, positive functional study or a reversible changes in the ECG consistent with ischemia). In subjects with coronary artery stenosis >75%, evidence of myocardial ischemia does not have to be documented

Exclusion Criteria

* Subject has a known hypersensitivity or contraindication to any of the following medications: heparin, aspirin, clopidogrel, prasugrel, ticagrelor, biolimus A9, everolimus, zotarolimus, stainless steel, cobalt chromium, contrast media (Patients with documented sensitivity to contrast media, which can be effectively premedicated with steroid and diphenhydramine may be enrolled. However, those with true anaphylaxis to prior contrast media should not be enrolled.)
* Subject in use of systemic (intravenous) biolimus A9, everolimus or zotarolimus within 12 months.
* Female subject of childbearing potential, unless a recent pregnancy test is negative, who possibly plans to become pregnant any time after enrollment into this study
* Subject planned an elective surgical procedure that would necessitate interruption of antiplatelet during the first 12 months post enrollment
* Subject with non-cardiac co-morbid condition with life expectancy < 2 year or that may result in protocol non-compliance (per site investigator's medical judgment)
* Subject with cardiogenic shock at presentation
* Subject who are actively participating in another drug or device investigational study, who have not completed the primary end point follow-up period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1960 (Actual)
Dates: Start 2013-01-16 (Actual); Primary Completion 2017-12-05 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Device-oriented composite | 24 months
  Device-oriented composite consisted of cardiac death, myocardial infarction not clearly attributable to a nontarget vessel, and clinically indicated target lesion revascularization (TLR) at 24-month clinical follow-up

SECONDARY OUTCOMES:
Patient-oriented composite | at 24 months
  Patient-oriented composite consisted of all-cause mortality, any myocardial infarction, and any revascularization at 24-month clinical follow-up
Device-oriented composite | 12 months
  Device-oriented composite at 12-month clinical follow-up
Patient-oriented composite | 12 months
  Patient-oriented composite at 12-month clinical follow-up
Each component of device- and patient-oriented composite | 12 months
  Each component of device- and patient-oriented composite at 12 months
Each component of device- and patient-oriented composite | 24 months
  Each component of device- and patient-oriented composite at 24 months
ARC defined stent thrombosis | 12 months
  ARC defined stent thrombosis at 12 months
ARC defined stent thrombosis | 24 months
  ARC defined stent thrombosis at 24 months
Stent thrombosis | 12 months
  ARC defined stent thrombosis at 12 months after randomization
Stent thrombosis | 24 months
  ARC defined stent thrombosis at 24 months after randomization
Bleeding complications defined by BARC definition | before discharge
  Bleeding complications defined by BARC definition before discharge

CONTACTS AND LOCATIONS:
Overall Officials: Junghan Yoon, M.D., Ph.D., Principal Investigator — Wonju Chrisitian Hospital
Locations (5):
- South Korea (5):
  - Wonju Christian Hospital, Wŏnju, Gangwon-do
  - Chonnam National University Hospital, Chuncheon
  - Daegu Catholic University Hospital, Daegu
  - Inha University Hospital, Incheon
  - Suncheon St. Carollo Hospital, Suncheon

REFERENCES:
- [Background] Kastrati A, Dibra A, Mehilli J, Mayer S, Pinieck S, Pache J, Dirschinger J, Schomig A. Predictive factors of restenosis after coronary implantation of sirolimus- or paclitaxel-eluting stents. Circulation. 2006 May 16;113(19):2293-300. doi: 10.1161/CIRCULATIONAHA.105.601823. Epub 2006 May 8. PMID 16682614
- [Background] Moses JW, Leon MB, Popma JJ, Fitzgerald PJ, Holmes DR, O'Shaughnessy C, Caputo RP, Kereiakes DJ, Williams DO, Teirstein PS, Jaeger JL, Kuntz RE; SIRIUS Investigators. Sirolimus-eluting stents versus standard stents in patients with stenosis in a native coronary artery. N Engl J Med. 2003 Oct 2;349(14):1315-23. doi: 10.1056/NEJMoa035071. PMID 14523139
- [Background] Pfisterer M, Brunner-La Rocca HP, Buser PT, Rickenbacher P, Hunziker P, Mueller C, Jeger R, Bader F, Osswald S, Kaiser C; BASKET-LATE Investigators. Late clinical events after clopidogrel discontinuation may limit the benefit of drug-eluting stents: an observational study of drug-eluting versus bare-metal stents. J Am Coll Cardiol. 2006 Dec 19;48(12):2584-91. doi: 10.1016/j.jacc.2006.10.026. Epub 2006 Nov 2. PMID 17174201
- [Background] Stone GW, Ellis SG, Cox DA, Hermiller J, O'Shaughnessy C, Mann JT, Turco M, Caputo R, Bergin P, Greenberg J, Popma JJ, Russell ME; TAXUS-IV Investigators. A polymer-based, paclitaxel-eluting stent in patients with coronary artery disease. N Engl J Med. 2004 Jan 15;350(3):221-31. doi: 10.1056/NEJMoa032441. PMID 14724301
- [Background] Holmes DR Jr, Kereiakes DJ, Laskey WK, Colombo A, Ellis SG, Henry TD, Popma JJ, Serruys PW, Kimura T, Williams DO, Windecker S, Krucoff MW. Thrombosis and drug-eluting stents: an objective appraisal. J Am Coll Cardiol. 2007 Jul 10;50(2):109-18. doi: 10.1016/j.jacc.2007.04.032. Epub 2007 May 22. PMID 17616294
- [Background] Iakovou I, Schmidt T, Bonizzoni E, Ge L, Sangiorgi GM, Stankovic G, Airoldi F, Chieffo A, Montorfano M, Carlino M, Michev I, Corvaja N, Briguori C, Gerckens U, Grube E, Colombo A. Incidence, predictors, and outcome of thrombosis after successful implantation of drug-eluting stents. JAMA. 2005 May 4;293(17):2126-30. doi: 10.1001/jama.293.17.2126. PMID 15870416
- [Background] Cutlip DE, Baim DS, Ho KK, Popma JJ, Lansky AJ, Cohen DJ, Carrozza JP Jr, Chauhan MS, Rodriguez O, Kuntz RE. Stent thrombosis in the modern era: a pooled analysis of multicenter coronary stent clinical trials. Circulation. 2001 Apr 17;103(15):1967-71. doi: 10.1161/01.cir.103.15.1967. PMID 11306525
- [Background] Doyle B, Rihal CS, O'Sullivan CJ, Lennon RJ, Wiste HJ, Bell M, Bresnahan J, Holmes DR Jr. Outcomes of stent thrombosis and restenosis during extended follow-up of patients treated with bare-metal coronary stents. Circulation. 2007 Nov 20;116(21):2391-8. doi: 10.1161/CIRCULATIONAHA.107.707331. Epub 2007 Nov 5. PMID 17984377
- [Background] Daemen J, Wenaweser P, Tsuchida K, Abrecht L, Vaina S, Morger C, Kukreja N, Juni P, Sianos G, Hellige G, van Domburg RT, Hess OM, Boersma E, Meier B, Windecker S, Serruys PW. Early and late coronary stent thrombosis of sirolimus-eluting and paclitaxel-eluting stents in routine clinical practice: data from a large two-institutional cohort study. Lancet. 2007 Feb 24;369(9562):667-78. doi: 10.1016/S0140-6736(07)60314-6. PMID 17321312
- [Background] Roukoz H, Bavry AA, Sarkees ML, Mood GR, Kumbhani DJ, Rabbat MG, Bhatt DL. Comprehensive meta-analysis on drug-eluting stents versus bare-metal stents during extended follow-up. Am J Med. 2009 Jun;122(6):581.e1-10. doi: 10.1016/j.amjmed.2008.12.019. PMID 19486720
- [Background] Kirtane AJ, Gupta A, Iyengar S, Moses JW, Leon MB, Applegate R, Brodie B, Hannan E, Harjai K, Jensen LO, Park SJ, Perry R, Racz M, Saia F, Tu JV, Waksman R, Lansky AJ, Mehran R, Stone GW. Safety and efficacy of drug-eluting and bare metal stents: comprehensive meta-analysis of randomized trials and observational studies. Circulation. 2009 Jun 30;119(25):3198-206. doi: 10.1161/CIRCULATIONAHA.108.826479. Epub 2009 Jun 15. PMID 19528338
- [Background] Mauri L, Hsieh WH, Massaro JM, Ho KK, D'Agostino R, Cutlip DE. Stent thrombosis in randomized clinical trials of drug-eluting stents. N Engl J Med. 2007 Mar 8;356(10):1020-9. doi: 10.1056/NEJMoa067731. Epub 2007 Feb 12. PMID 17296821
- [Background] Stone GW, Moses JW, Ellis SG, Schofer J, Dawkins KD, Morice MC, Colombo A, Schampaert E, Grube E, Kirtane AJ, Cutlip DE, Fahy M, Pocock SJ, Mehran R, Leon MB. Safety and efficacy of sirolimus- and paclitaxel-eluting coronary stents. N Engl J Med. 2007 Mar 8;356(10):998-1008. doi: 10.1056/NEJMoa067193. Epub 2007 Feb 12. PMID 17296824
- [Background] Caixeta A, Lansky AJ, Serruys PW, Hermiller JB, Ruygrok P, Onuma Y, Gordon P, Yaqub M, Miquel-Hebert K, Veldhof S, Sood P, Su X, Jonnavithula L, Sudhir K, Stone GW; SPIRIT II and III Investigators. Clinical follow-up 3 years after everolimus- and paclitaxel-eluting stents: a pooled analysis from the SPIRIT II (A Clinical Evaluation of the XIENCE V Everolimus Eluting Coronary Stent System in the Treatment of Patients With De Novo Native Coronary Artery Lesions) and SPIRIT III (A Clinical Evaluation of the Investigational Device XIENCE V Everolimus Eluting Coronary Stent System [EECSS] in the Treatment of Subjects With De Novo Native Coronary Artery Lesions) randomized trials. JACC Cardiovasc Interv. 2010 Dec;3(12):1220-8. doi: 10.1016/j.jcin.2010.07.017. PMID 21232715
- [Background] Kedhi E, Joesoef KS, McFadden E, Wassing J, van Mieghem C, Goedhart D, Smits PC. Second-generation everolimus-eluting and paclitaxel-eluting stents in real-life practice (COMPARE): a randomised trial. Lancet. 2010 Jan 16;375(9710):201-9. doi: 10.1016/S0140-6736(09)62127-9. Epub 2010 Jan 7. PMID 20060578
- [Background] Stone GW, Midei M, Newman W, Sanz M, Hermiller JB, Williams J, Farhat N, Mahaffey KW, Cutlip DE, Fitzgerald PJ, Sood P, Su X, Lansky AJ; SPIRIT III Investigators. Comparison of an everolimus-eluting stent and a paclitaxel-eluting stent in patients with coronary artery disease: a randomized trial. JAMA. 2008 Apr 23;299(16):1903-13. doi: 10.1001/jama.299.16.1903. PMID 18430909
- [Background] Stone GW, Rizvi A, Sudhir K, Newman W, Applegate RJ, Cannon LA, Maddux JT, Cutlip DE, Simonton CA, Sood P, Kereiakes DJ; SPIRIT IV Investigators. Randomized comparison of everolimus- and paclitaxel-eluting stents. 2-year follow-up from the SPIRIT (Clinical Evaluation of the XIENCE V Everolimus Eluting Coronary Stent System) IV trial. J Am Coll Cardiol. 2011 Jun 28;58(1):19-25. doi: 10.1016/j.jacc.2011.02.022. Epub 2011 Apr 21. PMID 21514084
- [Background] Serruys PW, Silber S, Garg S, van Geuns RJ, Richardt G, Buszman PE, Kelbaek H, van Boven AJ, Hofma SH, Linke A, Klauss V, Wijns W, Macaya C, Garot P, DiMario C, Manoharan G, Kornowski R, Ischinger T, Bartorelli A, Ronden J, Bressers M, Gobbens P, Negoita M, van Leeuwen F, Windecker S. Comparison of zotarolimus-eluting and everolimus-eluting coronary stents. N Engl J Med. 2010 Jul 8;363(2):136-46. doi: 10.1056/NEJMoa1004130. Epub 2010 Jun 16. PMID 20554978
- [Background] Silber S, Windecker S, Vranckx P, Serruys PW; RESOLUTE All Comers investigators. Unrestricted randomised use of two new generation drug-eluting coronary stents: 2-year patient-related versus stent-related outcomes from the RESOLUTE All Comers trial. Lancet. 2011 Apr 9;377(9773):1241-7. doi: 10.1016/S0140-6736(11)60395-4. Epub 2011 Apr 1. PMID 21459430
- [Background] Stefanini GG, Kalesan B, Serruys PW, Heg D, Buszman P, Linke A, Ischinger T, Klauss V, Eberli F, Wijns W, Morice MC, Di Mario C, Corti R, Antoni D, Sohn HY, Eerdmans P, van Es GA, Meier B, Windecker S, Juni P. Long-term clinical outcomes of biodegradable polymer biolimus-eluting stents versus durable polymer sirolimus-eluting stents in patients with coronary artery disease (LEADERS): 4 year follow-up of a randomised non-inferiority trial. Lancet. 2011 Dec 3;378(9807):1940-8. doi: 10.1016/S0140-6736(11)61672-3. Epub 2011 Nov 8. PMID 22075451
- [Background] Windecker S, Serruys PW, Wandel S, Buszman P, Trznadel S, Linke A, Lenk K, Ischinger T, Klauss V, Eberli F, Corti R, Wijns W, Morice MC, di Mario C, Davies S, van Geuns RJ, Eerdmans P, van Es GA, Meier B, Juni P. Biolimus-eluting stent with biodegradable polymer versus sirolimus-eluting stent with durable polymer for coronary revascularisation (LEADERS): a randomised non-inferiority trial. Lancet. 2008 Sep 27;372(9644):1163-73. doi: 10.1016/S0140-6736(08)61244-1. Epub 2008 Aug 31. PMID 18765162
- [Background] Luscher TF, Steffel J, Eberli FR, Joner M, Nakazawa G, Tanner FC, Virmani R. Drug-eluting stent and coronary thrombosis: biological mechanisms and clinical implications. Circulation. 2007 Feb 27;115(8):1051-8. doi: 10.1161/CIRCULATIONAHA.106.675934. PMID 17325255
- [Derived] Youn YJ, Lee JW, Ahn SG, Lee SH, Yoon J, Park KS, Lee JB, Yoo SY, Lim DS, Cho JH, Choi CU, Jeong MH, Han KR, Cha KS, Lee SY, Choi HH, Choi JW, Hyon MS, Kim MH. Randomized Comparison of Everolimus- and Zotarolimus-Eluting Coronary Stents With Biolimus-Eluting Stents in All-Comer Patients. Circ Cardiovasc Interv. 2020 Mar;13(3):e008525. doi: 10.1161/CIRCINTERVENTIONS.119.008525. Epub 2020 Mar 12. PMID 32160779
- [Derived] Youn YJ, Lee JW, Ahn SG, Lee SH, Choi HH, Choi H, Choi CU, Lee JB, Cho JH, Kang TS, Cho BR, Cha KS, Kim MH, Hyon MS, Cheong SS, Lim DS, Han KR, Jeong MH, Park KS, Yoon J. Study design and rationale of "a multicenter, open-labeled, randomized controlled trial comparing three 2nd-generation drug-eluting stents in real-world practice" (CHOICE trial). Am Heart J. 2013 Aug;166(2):224-9. doi: 10.1016/j.ahj.2013.04.014. Epub 2013 Jun 19. PMID 23895804